CLINICAL TRIAL: NCT04313244
Title: A Phase 3, Open-Label, Randomized Trial to Investigate the Immunogenicity and Safety of the Co-administration of a Subcutaneous Dengue Tetravalent Vaccine (Live, Attenuated) (TDV) and an Intramuscular Recombinant 9-Valent Human Papillomavirus (9vHPV) Vaccine in Subjects Aged ≥9 to <15 Years in an Endemic Country for Dengue
Brief Title: Immunogenicity and Safety of Dengue Tetravalent Vaccine (TDV) and Recombinant 9-valent Human Papillomavirus Vaccine (9vHPV) in Participants Aged ≥9 to <15 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DEN-308; 2022-003339-24 (EudraCT Number)
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Dengue Fever
Keywords: Drug therapy
MeSH Terms: conditions — Dengue | interventions — Dengue Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 9vHPV+TDV (Experimental): Participants will receive 0.5 mL 9vHPV intramuscularly (IM) with 0.5 mL TDV subcutaneously (SC) once on Day 1 (Month 0) followed by 0.5 mL TDV SC once on Day 90 (Month 3) and 0.5 mL 9vHPV IM once on Day 180 (Month 6).
  Interventions: Biological: 9vHPV Vaccine; Biological: Dengue Tetravalent Vaccine (TDV)
- 9vHPV (Experimental): Participants will receive 0.5 mL 9vHPV vaccine IM once on Day 1 (Month 0) followed by 0.5 mL 9vHPV vaccine IM once on Day 180 (Month 6).
  Interventions: Biological: 9vHPV Vaccine

INTERVENTIONS:
Biological: 9vHPV Vaccine — 9vHPV intramuscular injection
Biological: Dengue Tetravalent Vaccine (TDV) — TDV subcutaneous injection
  Other Names: TAK-003
  Arms: 9vHPV+TDV

SUMMARY:
The purpose of the study is to demonstrate the non-inferiority (NI) of the immune response to 2 doses of 9vHPV vaccine, 1 co-administered with TDV, compared with 2 doses of 9vHPV vaccine administered alone.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called Tetravalent Dengue Vaccine (TDV). The study will assess the immunogenicity and safety on the co-administration of 9vHPV vaccine with TDV in healthy participants aged ≥9 to <15 years.

The study will enroll approximately 614 healthy volunteers. Participants will be randomly assigned to one of the two treatment groups-

* Group 1
* Group 2

All participants will receive recombinant 9-valent Human Papillomavirus Vaccine (9vHPV) intramuscular (IM) in combination with Dengue Tetravalent Vaccine (TDV) subcutaneous (SC) injection on Day 1 (Month 0 ) followed by 9vHPV on Day 90 (Month 3) and TDV on Day 180 (Month 6) in Group 1. Participants will receive 9vHPV on Day 1 (Month 0) and Day 180 (Month 6) IM in Group 2.

This multi-center trial will be conducted in Thailand. The overall time to participate in this study is 12 months. Participants will make multiple visits to the clinic, after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs), and the clinical judgment of the investigator.
2. Participants who can comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. Has an elevated oral temperature ≥38°C (≥100.4°F) within 3 days of the intended date of vaccination.
2. Participants with contraindications, warnings and/or precautions to vaccination with Recombinant 9-valent Human Papillomavirus Vaccine (9vHPV) vaccine as specified within the prescribing information.
3. Has any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease.
4. Known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0) (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0).
   3. Administration of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (Month 0) or planned administration during the trial.
   4. Receipt of immunostimulants within 60 days prior to Day 1 (Month 0).
   5. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (Month 0).
   6. Human immunodeficiency virus (HIV) infection or HIV-related disease.
   7. Hepatitis B virus infection.
   8. Hepatitis C virus infection.
   9. Genetic immunodeficiency.
5. Abnormalities of splenic or thymic function.
6. Has a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
7. Who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of trial vaccine administration.
8. Who have used antipyretics and/or analgesic medications within 24 hours prior to vaccination. The reason for their use (prophylaxis versus treatment) must be documented. Trial entry should be delayed to allow for a full 24 hours to have passed since last use of antipyretics and/or analgesic medications.
9. Previous and planned vaccination (during the trial conduct), against any flavivirus (except Japanese encephalitis [JE]) including dengue, yellow fever (YF) viruses or tick-borne encephalitis.
10. Previous and planned vaccination (during the trial conduct) against HPV.
11. Previous participation in any clinical trial of a dengue or other flavivirus (eg, West Nile [WN] virus) candidate vaccine, except for participants who received placebo in those trials.
12. Has a current or previous infection with a flavivirus such as Zika, YF, JE, WN fever, tick-borne encephalitis or Murray Valley encephalitis.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 614 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (4):
- Thailand (4):
  - Siriraj Hospital, Bangkoknoi, Khet Bangkok Noi
  - King Chulalongkorn Memorial Hospital, Bangkok
  - The Hospital for Tropical Diseases, Bangkok
  - Thammasat University Hospital, Pathum Thani

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] El Hindi T, Anugulruengkitt S, Lapphra K, Limkittikul K, Tangsathapornpong A, Galindo CM, Hellwig M, Roubinis N, Schuring R, Biswal S, Folschweiller N. Immunogenicity and safety of the live-attenuated tetravalent dengue vaccine (TAK-003) co-administered with recombinant 9-valent human papillomavirus vaccine. Vaccine. 2025 Oct 24;65:127786. doi: 10.1016/j.vaccine.2025.127786. Epub 2025 Oct 6. PMID 41058426
- [Derived] El Hindi T, Anugulruengkitt S, Lapphra K, Limkittikul K, Tangsathapornpong A, Galindo-Tsoukas C, Hellwig M, Roubinis N, Schuring R, Biswal S, Folschweiller N. Immunogenicity and safety of the live-attenuated tetravalent dengue vaccine (TAK-003) co-administered with recombinant 9-valent human papillomavirus vaccine. Vaccine. 2025 Aug 30;62:127558. doi: 10.1016/j.vaccine.2025.127558. Epub 2025 Jul 31. PMID 40749348
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a399?idFilter=%5B%22C16021CSC%22%2C%22DEN-308%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in Thailand from 15 May 2021 to 19 July 2022.
Pre-assignment Details: Healthy participants aged ≥9 to <15 years in endemic areas for dengue were enrolled in this study to receive recombinant 9-valent human papillomavirus vaccine (9vHPV) alone or with tetravalent dengue vaccine (TDV).
Groups:
- 9vHPV+TDV: Participants received 0.5 mL 9vHPV intramuscularly (IM) and 0.5 mL TDV subcutaneously (SC) once on Day 1 (Month 0) followed by 0.5 mL TDV SC once on Day 90 (Month 3) and 0.5 mL 9vHPV IM once on Day 180 (Month 6).
- 9vHPV: Participants received 0.5 mL 9vHPV IM once on Day 1 (Month 0) followed by 0.5 mL 9vHPV IM once on Day 180 (Month 6).
Period: Overall Study
Arm/Group | 9vHPV+TDV | 9vHPV
Started | 307 | 307
Completed | 302 | 304
Not Completed | 5 | 3
Not completed — Withdrawal of Consent | 3 | 3
Not completed — Met Exclusion Criteria | 1 | 0
Not completed — Invalid Informed Consent Form (ICF) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized participants, regardless of whether any dose of the investigational products (IPs) was received.
Groups:
- 9vHPV+TDV: Participants received 0.5 mL 9vHPV IM and 0.5 mL TDV SC once on Day 1 (Month 0) followed by 0.5 mL TDV SC once on Day 90 (Month 3) and 0.5 mL 9vHPV IM once on Day 180 (Month 6).
- Total: Total of all reporting groups
Arm/Group | 9vHPV+TDV | 9vHPV | Total
Number analyzed (Participants) | 307 | 307 | 614
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (1.60) | 11.3 (1.59) | 11.2 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 156 | 306
  Male | 157 | 151 | 308
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 307 | 307 | 614
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 307 | 307 | 614
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 307 | 307 | 614
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number of participants analyzed is the number of participants with data available for height at the Baseline.
  centimeters (cm)
    number analyzed (Participants) | 306 | 307 | 613
    (all) | 147.68 (12.244) | 148.18 (11.374) | 147.93 (11.809)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: Number of participants analyzed is the number of participants with data available for weight at the Baseline.
  kilograms (kg)
    number analyzed (Participants) | 306 | 307 | 613
    (all) | 44.21 (15.913) | 44.37 (14.271) | 44.29 (15.101)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI=weight (kg) / [height (m)]^2 Population: Number of participants analyzed is the number of participants with data available for BMI at the Baseline.
  kilograms per meter square (kg/m^2)
    number analyzed (Participants) | 306 | 307 | 613
    (all) | 19.78 (4.912) | 19.88 (4.762) | 19.83 (4.834)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) for Human Papillomavirus (HPV) Types 6, 11, 16, 18, 31, 33, 45, 52, 58
Description: GMTs for HPV were measured by immunoglobulin G binding assay (IgGBA) assay. HPV-6, HPV-11, HPV-16, HPV-18, HPV-31, HPV-33, HPV-45, HPV-52 and HPV-58 were the types of HPV analyzed.
Time Frame: Day 210 (Month 7)
Population: The Per-protocol Set (PPS) excluded all participants seropositive to any HPV type at Baseline and included all participants from the Full Analysis Set (FAS) who had no major protocol violations. Overall number of participants analyzed is the number of participants available for analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 9vHPV+TDV | 9vHPV
Number analyzed (Participants) | 237 | 234
titer
  HPV-6 | 1633.693 [1465.31 to 1821.43] | 1790.986 [1556.08 to 2061.35]
  HPV-11 | 1342.745 [1225.64 to 1471.04] | 1325.192 [1164.58 to 1507.95]
  HPV-16 | 7777.694 [6989.76 to 8654.45] | 7822.564 [6701.83 to 9130.71]
  HPV-18 | 2309.629 [2075.91 to 2569.66] | 2506.309 [2182.67 to 2877.93]
  HPV-31 | 1690.941 [1529.39 to 1869.55] | 1736.943 [1515.05 to 1991.33]
  HPV-33 | 1138.716 [1019.66 to 1271.67] | 1179.469 [1033.66 to 1345.84]
  HPV-45 | 504.033 [453.46 to 560.24] | 584.198 [509.91 to 669.31]
  HPV-52 | 585.606 [533.44 to 642.87] | 561.007 [492.77 to 638.69]
  HPV-58 | 1163.600 [1060.23 to 1277.05] | 1284.504 [1130.63 to 1459.32]

2. Secondary Outcome: Percentage of Participants With Seropositivity for HPV Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 as Measured by Immunoglobulin G Binding Assay (IgGBA)
Description: Seropositive for HPV is defined as anti-HPV titers greater or equal to the prespecified cutoffs for any of the 9 HPV serotypes: HPV-6, HPV-11, HPV-16, HPV-18, HPV-31, HPV-33, HPV-45, HPV-52 and HPV-58, measured by IgGBA. The serostatus cut-off is the antibody titer level above the assay's lower limit of quantification that reliably distinguishes sera samples classified by clinical likelihood of HPV infection and positive or negative status by previous versions of IgGBA or equivalent assay. The serostatus cut-offs for the 9 HPV serotypes: HPV-6= 9, HPV-11= 6, HPV-16= 5, HPV-18= 5, HPV-31= 3, HPV-33= 4, HPV-45= 3, HPV-52= 5 and HPV-58= 5. Percentages are rounded off to the nearest decimal point.
Time Frame: Day 210 (Month 7)
Population: The PPS excluded all participants seropositive to any HPV type at Baseline and included all participants from the FAS who had no major protocol violations. Overall number of participants analyzed is the number of participants available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 9vHPV+TDV | 9vHPV
Number analyzed (Participants) | 237 | 234
percentage of participants
  HPV-6 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]
  HPV-11 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]
  HPV-16 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]
  HPV-18 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]
  HPV-31 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]
  HPV-33 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]
  HPV-45 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]
  HPV-52 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]
  HPV-58 | 100.0 [98.5 to 100.0] | 99.1 [96.9 to 99.9]

3. Secondary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes
Description: GMTs of neutralizing antibodies for each of the 4 dengue serotypes were measured by microneutralization test 50% (MNT50). The four dengue serotypes: DENV-1, DENV-2, DENV-3 and DENV-4. As prespecified in the protocol, the data for this outcome measure was collected and analyzed for participants in the 9vHPV+TDV arm group only.
Time Frame: Day 120 (Month 4)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 9vHPV+TDV
Number analyzed (Participants) | 238
titer
  DENV-1 | 719.1 [577.8 to 895.0]
  DENV-2 | 1691.4 [1411.0 to 2027.4]
  DENV-3 | 555.4 [462.8 to 666.6]
  DENV-4 | 494.3 [420.8 to 580.6]

4. Secondary Outcome: Percentage of Participants With Seropositivity for Each of the 4 Dengue Serotypes
Description: Seropositivity is defined as a reciprocal neutralizing antibody titer ≥10 for any of the 4 dengue serotypes. The four dengue serotypes: DENV-1, DENV-2, DENV-3 and DENV-4. As prespecified in the protocol, the data for this outcome measure was collected and analyzed for participants in the 9vHPV+TDV arm group only. Percentages are rounded off to the nearest decimal point.
Time Frame: Day 120 (Month 4)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 9vHPV+TDV
Number analyzed (Participants) | 238
percentage of participants
  DENV-1 | 100.0 [98.5 to 100.0]
  DENV-2 | 99.6 [97.7 to 100.0]
  DENV-3 | 100.0 [98.5 to 100.0]
  DENV-4 | 100.0 [98.5 to 100.0]

5. Secondary Outcome: Percentage of Participants With Seropositivity for Multiple (2, 3 or 4) Dengue Serotypes
Description: Seropositivity is defined as a reciprocal neutralizing antibody titer ≥10 for any of the 4 dengue serotypes. The dengue virus serotypes are DENV-1, DENV-2, DENV-3 and DENV-4. Seropositive for multiple dengue serotypes were summarized for categories with at least one participant with event: trivalent (seropositive for 3 dengue serotypes), and tetravalent (seropositive for all 4 dengue serotypes). As prespecified in the protocol, the data for this outcome measure was collected and analyzed for participants in the 9vHPV+TDV arm group only. Percentages are rounded off to the nearest decimal point.
Time Frame: Day 120 (Month 4)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 9vHPV+TDV
Number analyzed (Participants) | 238
percentage of participants
  Trivalent | 0.4 [0.0 to 2.3]
  Tetravalent | 99.6 [97.7 to 100.0]

6. Secondary Outcome: Percentage of Participants With Solicited Local Adverse Events for 7 Days Following Vaccination by Severity
Description: Solicited local adverse events (AEs) (at injection site) were collected by participants using diary cards within 7 days after vaccination and included: Pain [Grade 0 (no pain), 1 (mild: no interference with daily activity), 2 (moderate: interference with daily activity with or without treatment) and 3 (severe: prevents daily activity with or without treatment)]; erythema and swelling [Grade 0 (<25 millimeters [mm]), 1 (25 - ≤ 50 mm), 2 (>50 - ≤ 100 mm), 3 (> 100 mm)]. Percentages are rounded off to the nearest decimal point. The data for solicited local adverse events after any vaccination are presented. Only those categories with at least 1 participant with event are reported.
Time Frame: Up to 7 days (Day of vaccination + 6 subsequent days) after each vaccination
Population: Safety Set included all randomized participants who received at least 1 dose of IPs.
Measure: Number; unit: percentage of participants
Arm/Group | 9vHPV+TDV | 9vHPV
Number analyzed (Participants) | 307 | 307
percentage of participants
  Pain: Mild | 54.1 | 42.8
  Pain: Moderate | 9.5 | 6.5
  Pain: Severe | 0.7 | 0
  Erythema: Mild | 7.5 | 0
  Erythema: Moderate | 0.7 | 0
  Swelling: Mild | 3.3 | 0

7. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) for 14 Days Following Vaccination by Severity
Description: Solicited systemic AEs were collected by participants using diary cards within 14 days after vaccination and included fever, headache, asthenia, malaise, and myalgia. Severity grades were: Grade 0: none, Grade 1: mild (no interference with daily activity), Grade 2: moderate (interference with daily activity with or without treatment), Grade 3: severe (prevents normal daily activity with or without treatment). Fever is defined as body temperature greater than or equal to 38°C (100.4 degrees Fahrenheit [°F]). Only categories with at least one participant with event following any vaccination are reported. Percentages are rounded off to the nearest decimal point. The data for solicited systemic adverse events after any vaccination are presented.
Time Frame: Up to 14 days (Day of vaccination + 13 subsequent days) after each vaccination
Population: Safety Set included all randomized participants who received at least 1 dose of IPs.
Measure: Number; unit: percentage of participants
Arm/Group | 9vHPV+TDV | 9vHPV
Number analyzed (Participants) | 307 | 307
percentage of participants
  Headache: Mild | 20.0 | 18.0
  Headache: Moderate | 3.0 | 0.7
  Headache: Severe | 0.3 | 0
  Asthenia: Mild | 16.7 | 12.1
  Asthenia: Moderate | 2.0 | 1.0
  Asthenia: Severe | 0.3 | 0
  Malaise: Mild | 17.7 | 10.5
  Malaise: Moderate | 2.0 | 1.3
  Malaise: Severe | 0.3 | 0
  Myalgia: Mild | 36.1 | 27.8
  Myalgia: Moderate | 7.9 | 2.3
  Myalgia: Severe | 0.3 | 0.3
  Fever: 38.0°C to <38.5°C | 2.0 | 0.3
  Fever: 38.5°C to <39.0°C | 0.3 | 0
  Fever: 39.0°C to <39.5°C | 0.3 | 0

8. Secondary Outcome: Percentage of Participants With Any Unsolicited AEs for 28 Days Following Vaccination
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a study vaccine; it does not necessarily have to have a causal relationship with study vaccine administration. Percentages are rounded off to the nearest decimal point. The data for unsolicited adverse events after any vaccination are presented.
Time Frame: Up to 28 days (Day of vaccination + 27 subsequent days) after each vaccination
Population: Safety Set included all randomized participants who received at least 1 dose of IPs.
Measure: Number; unit: percentage of participants
Arm/Group | 9vHPV+TDV | 9vHPV
Number analyzed (Participants) | 307 | 307
percentage of participants | 8.8 | 2.6

9. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence or effect that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important which may require intervention to prevent the items listed above or may expose the participant to danger.
Time Frame: From first vaccination (Day 1 [Month 0]) through end of study (Day 360 [Month 12])
Population: Safety Set included all randomized participants who received at least 1 dose of IPs.
Measure: Number; unit: percentage of participants
Arm/Group | 9vHPV+TDV | 9vHPV
Number analyzed (Participants) | 307 | 307
percentage of participants | 10.1 | 7.2

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events: From first vaccination (Day 1 [Month 0]) through end of study (Day 360 [Month 12]); Non-serious adverse events: Up to 28 days (day of vaccination + 27 days) after each vaccination
Description: Safety Set included all randomized participants who received at least 1 dose of IPs.
Arm/Group | 9vHPV+TDV | 9vHPV
All-Cause Mortality (participants affected / at risk) | 0/307 | 0/307
Serious Adverse Events (participants affected / at risk) | 31/307 | 22/307
Other Adverse Events (participants affected / at risk) | 253/307 | 223/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 9vHPV+TDV (N=307) | 9vHPV (N=307)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 26 | 19
COVID-19 pneumonia (Infections and infestations) | 2 | 2
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 9vHPV+TDV (N=307) | 9vHPV (N=307)
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 58 | 40
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 92 | 57
Fever (General disorders) | 8 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 71 | 59
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Malaise (General disorders) | 62 | 36
Myalgia (Musculoskeletal and connective tissue disorders) | 135 | 93
Nasopharyngitis (Infections and infestations) | 3 | 0
Pain (General disorders) | 225 | 184
Pyrexia (General disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Swelling (General disorders) | 64 | 52
Syncope (Nervous system disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT04313244/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT04313244/SAP_001.pdf